CLINICAL TRIAL: NCT03705052
Title: Patient's and Caregiver's Expectations and Preferences Concerning Art Therapy Activities for Cancer Support in Light of Founding an Art Therapy Centre
Brief Title: Patient's and Caregiver's Expectations and Preferences Concerning Art Therapy Activities for Cancer Support
Acronym: PREFERENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Principal investigator, General Hospital Groeninge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AZGS2018026
Record Dates: First submitted 2018-09-24; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Psychological Distress
Keywords: Art therapy; surveys and questionnaires; patient; caregiver
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Patients and caregivers were asked to complete a questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients and caregivers were asked to complete a questionnaire

SUMMARY:
Cancer patients and their caregivers often experience difficulties in coping with the cancer diagnosis and the treatment that follows. Creative art therapy could support cancer patients and their caregivers in coping with these issues by using their creativity and self-expression. The aim of this study for the investigator's research team is to create a clear image of what cancer patients and their caregivers expect of supportive care to help them coping with cancer diagnosis, cancer therapy and life after cancer. This is a prospective, interventional study. Cancer patients and their caregivers will be approached to participate in this study. They will be asked to complete a questionnaire about their satisfaction with the current support they get to help them coping with cancer diagnosis, cancer therapy and life after cancer and whether they would like to participate in an art therapy program, which art therapy forms they would like to participate in, how they would like them to be organized, etc.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking patients and caregivers
* Patients and caregivers presenting at the outpatient clinic, including the day-care clinic and follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Response rate | At study inclusion

SECONDARY OUTCOMES:
Activities of interest assessed by questionnary | At study inclusion
Preference on organization of activities evaluated by questionnary | At study inclusion
Patient or caregiver characteristics (sex, age, diagnosis) collected by questionnary | At study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philip Derbuyne, MD, PhD, MSc, FRCP, Principal Investigator — General Hospital Groeninge
Locations (1):
- General Hospital Groeninge, Cancer Center, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visser A, Op 't Hoog M. Education of creative art therapy to cancer patients: evaluation and effects. J Cancer Educ. 2008;23(2):80-4. doi: 10.1080/08858190701821204. PMID 18569242
- [Background] Geue K, Goetze H, Buttstaedt M, Kleinert E, Richter D, Singer S. An overview of art therapy interventions for cancer patients and the results of research. Complement Ther Med. 2010 Jun-Aug;18(3-4):160-70. doi: 10.1016/j.ctim.2010.04.001. Epub 2010 May 15. PMID 20688262
- [Background] Bar-Sela G, Atid L, Danos S, Gabay N, Epelbaum R. Art therapy improved depression and influenced fatigue levels in cancer patients on chemotherapy. Psychooncology. 2007 Nov;16(11):980-4. doi: 10.1002/pon.1175. PMID 17351987
- [Background] Walsh SM, Martin SC, Schmidt LA. Testing the efficacy of a creative-arts intervention with family caregivers of patients with cancer. J Nurs Scholarsh. 2004;36(3):214-9. doi: 10.1111/j.1547-5069.2004.04040.x. PMID 15495489